CLINICAL TRIAL: NCT05173259
Title: Effect of Side Switch Frequency on Masticatory Mixing Ability and Perception of Taste, Muscular Fatigue and Saliva Production: A Randomized Crossover Trial.
Brief Title: Masticatory Side-switch and Mixing Ability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Jordi Martinez-Gomis, Associate Professor DDS. PhD, University of Barcelona
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HOUB 44/2021
Record Dates: First submitted 2021-12-27; First posted 2021-12-29 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Chewing Problem; Mastication Disorder
Keywords: Chewing side; Masticatory side-switch; Mastication; Masticatory rhythm; Masticatory performance; Masticatory mixing ability
MeSH Terms: interventions — RBM5 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- F-R/L-G05/G15/G25 or G25/G15/G05-L/R-F Sequence (Active Comparator): First, 2 freestyle masticatory assays (F). Second, 2 only-right (R) and 2 only-left (L) masticatory assays in the following order (R-L-L-R). Third, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G05-G15-G25-G25-G15-G05).
  Or
  First, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G05-G15-G25-G25-G15-G05). Second, 2 only-left (L) and 2 only-right (R) masticatory assays in the following order (L-R-R-L). Third, 2 freestyle masticatory assays (F).
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: G05; Behavioral: G15; Behavioral: G25
- F-R/L-G05/G25/G15 or G15/G25/G05-F-L/R Sequence (Active Comparator): First, 2 freestyle masticatory assays (F). Second, 2 only-right (R) and 2 only-left (L) masticatory assays in the following order (R-L-L-R). Third, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G05-G25-G15-G15-G25-G05).
  Or
  First, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G05-G25-G15-G15-G25-G05). Second, 2 only-left (L) and 2 only-right (R) masticatory assays in the following order (L-R-R-L). Third, 2 freestyle masticatory assays (F).
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: G05; Behavioral: G15; Behavioral: G25
- F-R/L-G15/G05/G25 or G25/G05/G15-F-L/R Sequence (Active Comparator): First, 2 freestyle masticatory assays (F). Second, 2 only-right (R) and 2 only-left (L) masticatory assays in the following order (R-L-L-R). Third, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G05-G15-G25-G25-G15-G05).
  Or
  First, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G15-G05-G25-G25-G05-G15). Second, 2 only-left (L) and 2 only-right (R) masticatory assays in the following order (L-R-R-L). Third, 2 freestyle masticatory assays (F).
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: G05; Behavioral: G15; Behavioral: G25
- F-R/L-G15/G25/G05 or G05/G25/G15-F-L/R Sequence (Active Comparator): First, 2 freestyle masticatory assays (F). Second, 2 only-right (R) and 2 only-left (L) masticatory assays in the following order (R-L-L-R). Third, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G15-G25-G05-G05-G25-G15).
  Or
  First, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G15-G25-G05-G05-G25-G15). Second, 2 only-left (L) and 2 only-right (R) masticatory assays in the following order (L-R-R-L). Third, 2 freestyle masticatory assays (F).
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: G05; Behavioral: G15; Behavioral: G25
- F-R/L-G25/G05/G15 or G15/G05/G25-F-L/R Sequence (Active Comparator): First, 2 freestyle masticatory assays (F). Second, 2 only-right (R) and 2 only-left (L) masticatory assays in the following order (R-L-L-R). Third, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G25-G05-G15-G15-G05-G25).
  Or
  First, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G25-G05-G15-G15-G05-G25). Second, 2 only-left (L) and 2 only-right (R) masticatory assays in the following order (L-R-R-L). Third, 2 freestyle masticatory assays (F).
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: G05; Behavioral: G15; Behavioral: G25
- F-R/L-G25/G15/G05 or G05/G15/G25-F-L/R Sequence (Active Comparator): First, 2 freestyle masticatory assays (F). Second, 2 only-right (R) and 2 only-left (L) masticatory assays in the following order (R-L-L-R). Third, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G25-G15-G05-G05-G15-G25).
  Or
  First, 6 masticatory assays changing in 5% (G05), 15% (G15) or 25% (G25) in the following order (G25-G15-G05-G05-G15-G25). Second, 2 only-left (L) and 2 only-right (R) masticatory assays in the following order (L-R-R-L). Third, 2 freestyle masticatory assays (F).
  Interventions: Behavioral: F; Behavioral: R; Behavioral: L; Behavioral: G05; Behavioral: G15; Behavioral: G25

INTERVENTIONS:
Behavioral: F — The participant will be asked to chew the two-coloured chewing gum naturally.
Behavioral: R — The participant will be asked to chew the two-coloured chewing gum on the right-side.
Behavioral: L — The participant will be asked to chew the two-coloured chewing gum on the left-side.
Behavioral: G05 — The participant will be asked to chew the two-coloured chewing gum changing the side in 5%.
Behavioral: G15 — The participant will be asked to chew the two-coloured chewing gum changing the side in 15%.
Behavioral: G25 — The participant will be asked to chew the two-coloured chewing gum changing the side in 25%.

SUMMARY:
The main aim of this cross-over intervention study is to assess the effect of masticatory side-switch frequency on different aspects of masticatory function, including masticatory mixing ability and rhythm. A secondary aim is to explore the subjective perception of taste, muscular fatigue, and saliva production through a VAS. Thirty-six volunteers recruited for convenience, among students of the Degree of Dentistry of the Faculty of Medicine and Health Sciences of the University of Barcelona, will perform 6 tests, each consisting of 2 assays, chewing a two-coloured chewing gum, during 40 masticatory cycles. The tests will be randomised masticatory sequences of "free-style", "unilateral-right", "unilateral-left", switching the chewing side at 5% "G05", at 15% "G15" and at 25% "G25". Video recordings of these tests will be made to later assess, on slow playback, the change of the chewing side and the masticatory rhythm. The masticatory mixing ability will be determined through the scanning and posterior analysis of the red-channel in the histogram plug-in in "ImageJ" (R).

DETAILED DESCRIPTION:
This this cross-over intervention study aims to assess the effect of masticatory side-switch frequency on different objective aspects of masticatory function, including masticatory mixing ability and rhythm, as well as the subjective perception of taste, muscular fatigue, and saliva production through a VAS. Each of the thirty-six volunteers recruited for convenience, among students of the Degree of Dentistry of the Faculty of Medicine and Health Sciences of the University of Barcelona, will perform 6 tests, each consisting of 2 assays, chewing a two-coloured chewing gum, during 40 masticatory cycles. One test involves freestyle mastication in which the participant will be asked to masticate the chewing gum. Two tests involve chewing the gum unilaterally (i.e., only on the right-hand side, and only on the left) varying the order of these assays. In the last three tests, the volunteer will switch chewing side in 5% (G05), 15% (G15), or 25% (G25) respectively; the sequence of the assays will be randomized. Twenty-four of these volunteers will be randomly selected to repeat these tests after a period of two weeks. The masticatory mixing ability will be determined through the "mixing capacity index" (MCI), obtained from through the scanning and posterior analysis of the red-channel in the histogram plug-in in "ImageJ" (R), and the masticatory rhythm will be assessed through the masticatory frequency as the ratio of masticatory cycle number to masticatory time. The control variables will include age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Natural dentition (minimum 24 teeth)

Exclusion Criteria:

* Active orthodontics treatment.
* Intraoral pain.
* Temporomandibular joint pain.
* Masticatory muscle pain.
* Large dental restorations.
* Dental prosthesis.
* Edentulous spaces.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Masticatory mixing ability | 1 hour
  Masticatory mixing ability will be calculated from the mixing capacity for each type of test (free, right, left and guided). Chewing gum will flattened between two rigid surfaces to a thickness of 1.5 mm. The two sides of the chewing gum will then be scanned at a resolution of 300 dpi. The images will be processed with "ImageJ" with the "Color-Histogram" plugin. Before mixing, the green and red color of the chewing gum are represented in the histogram of the red channel as two separate peaks: one in low intensity and one in high intensity, representing the green and red color of chewing gum, respectively. After mixing, the colors are mixed and so the two peaks merge into one peak. The standard deviation of the intensity distribution is taken as a measure of the mixture of the two colors in the chewing gum. The standard deviation at an early stage of mixing is relatively high, and decreases as the colors are mixed; thus, a high value of the mixing index means a high mixing capacity.
Side-switch Index | 1 hour
  The number of side switches during the 40 masticatory cycles for each assay will be determined using slow playback of the video recordings of the freestyle mastication test. In the case that this switch is a change of side from left to right or right to left, we will assign a value of "1". If this switch consists of a change from the right or left to central or vice versa, we will assign a value of "0.5". If there is no change of side, the value assigned to this chewing cycle will be "0". To determine the Side-switch Index, the number of side changes will be divided by the maximum number of changes possible during these 5 assays (78).

SECONDARY OUTCOMES:
Masticatory Frequency | 1 hour
  Masticatory frequency will be assessed as the ratio of masticatory cycle number to masticatory time (in cycles per minute).
Degree of muscular fatigue during this masticatory assay | 1 hour
  The degree of muscular fatigue while chewed the gum was assessed by asking the question "How much muscular fatigue do you think this masticatory test caused you?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Participants will rate the masticatory test after each assay.
Degree of salivary secretion during this masticatory assay | 1 hour
  The degree of salivary secretion while chewed the gum was assessed by asking the question "How much saliva secretion do you think this masticatory test caused you?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Participants will rate the masticatory test after each assay.
Degree of taste perception during this masticatory assay | 1 hour
  The degree of taste perception while chewed the gum was assessed by asking the question "To what degree do you think this masticatory test facilitates taste perception?" using a 0-10 point scale (considering 0= Not at all to 10= very much). Participants will rate the masticatory test after each assay.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, University of Barcelona, L'Hospitalet de Llobregat, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Bilt A. Assessment of mastication with implications for oral rehabilitation: a review. J Oral Rehabil. 2011 Oct;38(10):754-80. doi: 10.1111/j.1365-2842.2010.02197.x. Epub 2011 Jan 17. PMID 21241351
- [Background] van der Bilt A, Abbink JH. The influence of food consistency on chewing rate and muscular work. Arch Oral Biol. 2017 Nov;83:105-110. doi: 10.1016/j.archoralbio.2017.07.011. Epub 2017 Jul 20. PMID 28750270
- [Background] Mizumori T, Tsubakimoto T, Iwasaki M, Nakamura T. Masticatory laterality--evaluation and influence of food texture. J Oral Rehabil. 2003 Oct;30(10):995-9. doi: 10.1046/j.1365-2842.2003.01086.x. PMID 12974859
- [Background] Flores-Orozco EI, Rovira-Lastra B, Peraire M, Salsench J, Martinez-Gomis J. Reliability of a visual analog scale for determining the preferred mastication side. J Prosthet Dent. 2016 Feb;115(2):203-8. doi: 10.1016/j.prosdent.2015.07.006. Epub 2015 Oct 9. PMID 26455536
- [Background] Mioche L, Hiiemae KM, Palmer JB. A postero-anterior videofluorographic study of the intra-oral management of food in man. Arch Oral Biol. 2002 Apr;47(4):267-80. doi: 10.1016/s0003-9969(02)00007-9. PMID 11922870
- [Background] Woda A, Foster K, Mishellany A, Peyron MA. Adaptation of healthy mastication to factors pertaining to the individual or to the food. Physiol Behav. 2006 Aug 30;89(1):28-35. doi: 10.1016/j.physbeh.2006.02.013. Epub 2006 Apr 3. PMID 16581096
- [Background] Remijn L, Groen BE, Speyer R, van Limbeek J, Nijhuis-van der Sanden MW. Reproducibility of 3D kinematics and surface electromyography measurements of mastication. Physiol Behav. 2016 Mar 1;155:112-21. doi: 10.1016/j.physbeh.2015.11.018. Epub 2015 Nov 23. PMID 26617403
- [Background] Mizumori T, Arai K. Tsubakimoto T, Yatani H. Chewing side continuity and masticatory performance. Prosthodont Res Pract 2006;5:10-4.
- [Background] Weijenberg RA, Scherder EJ, Visscher CM, Gorissen T, Yoshida E, Lobbezoo F. Two-colour chewing gum mixing ability: digitalisation and spatial heterogeneity analysis. J Oral Rehabil. 2013 Oct;40(10):737-43. doi: 10.1111/joor.12090. Epub 2013 Aug 9. PMID 23927753
- [Background] van der Bilt A, Speksnijder CM, de Liz Pocztaruk R, Abbink JH. Digital image processing versus visual assessment of chewed two-colour wax in mixing ability tests. J Oral Rehabil. 2012 Jan;39(1):11-7. doi: 10.1111/j.1365-2842.2011.02229.x. Epub 2011 Jun 27. PMID 21707695
- [Background] Schimmel M, Christou P, Miyazaki H, Halazonetis D, Herrmann FR, Muller F. A novel colourimetric technique to assess chewing function using two-coloured specimens: Validation and application. J Dent. 2015 Aug;43(8):955-64. doi: 10.1016/j.jdent.2015.06.003. Epub 2015 Jun 22. PMID 26111925
- [Background] Montero J, Leiva LA, Martin-Quintero I, Barrios-Rodriguez R. Chewing Performance Calculator: An interactive clinical method for quantifying masticatory performance. J Prosthet Dent. 2021 Jan;125(1):82-88. doi: 10.1016/j.prosdent.2019.10.006. Epub 2020 Jan 25. PMID 31987585
- [Background] Yousof Y, Salleh NM, Yusof F. Quantitative Evaluation of Masticatory Performance with Two-Color Mixing Ability Test: Development of a New Digital Method. Int J Prosthodont. 2020 Mar/Apr;33(2):224-228. doi: 10.11607/ijp.6568. PMID 32069348
- [Background] van der Bilt A, Mojet J, Tekamp FA, Abbink JH. Comparing masticatory performance and mixing ability. J Oral Rehabil. 2010 Feb;37(2):79-84. doi: 10.1111/j.1365-2842.2009.02040.x. Epub 2009 Dec 7. PMID 19968766